CLINICAL TRIAL: NCT04427891
Title: Study of Changes in Abdominal Fluid in Connection With Peritonitis. A Descriptive Study in Patients With Purulent or Fecal Peritonitis.
Brief Title: Characteristics of Abdominal Fluid in Patients With Diverticulitis Hinchey III or IV
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Eva Haglind, MD, PhD, professor, professor, Sahlgrenska University Hospital
Other Study IDs: 2019-06114
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Perforated Diverticulitis
Keywords: perforated diverticulitis; peritonitis; protein changes; microbiota
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — periferal blood, abdominal fluid, colon wall, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group I: Patients undergoing emergency surgery due to perforated diverticulitis with peritonitis.
  No intervention, samples from abdominal fluid, blood, tissue, feces
- Group II: Patients with colorectal cancer undergoing elective surgery. No intervention. Samples as for Group I
- Group III: Patients with mild diverticulitis, not undergoing surgery. No intervention. Samples from blood and feces.

SUMMARY:
Perforated diverticulitis of the colon can be complicated by peritonitis, either purulent or fecal. Both are life threatening conditions requiring emergency surgery. The background in terms of reasons for inflammation (diverticulitis) and perforation to develop is unknown. In this study we focus on specific changes associated with inflammation, both in tissues and of fecal and mucosal microbiota.

DETAILED DESCRIPTION:
A prospective study of abdominal fluid, periferal blood, tissues as well as feces in Patients (perforated diverticulitis with peritonitis undergoing emergency surgery, Group I), and in Controls (patients operated due to colorectal cancer, Group II; patients with mild diverticulitis not needing surgery, Group III).

Immune acitvity in abdominal fluid and periferal blood by immunoassay of 92 individual proteins. mRNA expression of 96 specific genes in tissue samples. Quatification of bacterial diversity in feces and colon mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Signs of perforated diverticulitis with peritonitis and decision to perform emergency surgery (Group I)
* Signs of acute diverticulitis and no decision of emergency surgery (Group II)
* Patients with colorectal cancer planned for elective surgery (Group III)

Exclusion Criteria:

* No surgery performed (Group I and III)
* Withdrawn consent (any group)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The aim is to study immune responses in patients with perforated divrticulitis leading to peritonitis and emergency surgery. This group will be compared with patients operated for colorectal cancer and patients with uncomplicated (mild) diverticulitis not undergoing surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
inflammatory response | index surgery (Groups I and II)/ emergency room (Group III)
  determination of levels of 92 proteins in abdominal fluid and blood

SECONDARY OUTCOMES:
inflammatory response in tissue | index surgery (Groups I and II)/ emergency room (Group III)
  RNA sequencing (96 spcific genes) in abdominal tissue
microbiota composition | index surgery (Groups I and II)/ emergency room (Group III)
  PCR amplification, cloning and sequencing of genes

CONTACTS AND LOCATIONS:
Overall Officials: Eva Haglind, MD,PhD, Principal Investigator — Sahlgrenska univesitetssjukhuset
Locations (1):
- Sahlgrenska University Hospital/Östra, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No